CLINICAL TRIAL: NCT00234221
Title: Services Interventions for Injured ED Problem Drinkers
Brief Title: Project Health Link: Connecting Patients With Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Frederic C. Blow, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01AA014665-01A1 (NIH)
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Strengths Based Case Management Model (SBCM) (Active Comparator): The Strengths Based Case Management Model (SBCM) consists of 5 case-management sessions designed to promote linkage and engagement in assessment and treatment services, while assisting with the patient's perceived needs, as well as personal strengths and barriers to linkage and engagement.
  Interventions: Behavioral: Strengths Based Case Management
- Motivational Enhancement Therapy (MET) (Active Comparator): The MET therapist will conduct 2 motivational enhancement sessions to work through the content of an educational workbook targeting the participant's alcohol use/abuse with the goal of negotiating a 'contract' to: 1) link to services, with the eventual goal of seeking and receiving specialized alcohol treatment; or 2) provide a strategy to self-monitor alcohol use, consider consequences, and later seek assessment.
  Interventions: Behavioral: Motivational Enhancement Therapy
- Brief Informational Feedback (BIF) session (Active Comparator): Subjects will receive brief informational feedback on the results of their alcohol screening and assessment and encouragement to seek treatment.
  Interventions: Behavioral: Brief Informational Feedback

INTERVENTIONS:
Behavioral: Strengths Based Case Management
  Arms: Strengths Based Case Management Model (SBCM)
Behavioral: Motivational Enhancement Therapy
  Arms: Motivational Enhancement Therapy (MET)
Behavioral: Brief Informational Feedback
  Arms: Brief Informational Feedback (BIF) session

SUMMARY:
This study will compare three alternative interventions in the emergency department (ED) to promote substance abuse assessment, referral, and treatment entry: 1) a 5 session strengths-based case management model (SBCM); 2) a 2-session motivational enhancement therapy (MET); or 3) a one-time brief informational feedback (BIF) session. The primary outcome variables for this trial include follow-through on receiving an assessment and referral, and treatment engagement. Additional outcomes include degree of treatment completion, alcohol-related measures, health service utilization, health status changes, and psychosocial factors.

ELIGIBILITY:
Inclusion Criteria:

* (1) adults age 19 - 60 presenting to the Emergency Department at Hurley Medical Center within 24 hours of an injury; (2) ability to provide informed consent.

For intervention portion of the project: (1) meets DSM-IV criteria for alcohol abuse or dependence in the following year. (Patients who meet abuse/dependence criteria for alcohol may also be using other drugs. They will be included in the study only if they do not meet criteria for past year drug abuse/dependence).

Exclusion Criteria:

* (1) adult patients who do not understand English; (2) prisoners; (3) pregnant women; (4) institutionalized patients (e.g. nursing home residents); (5) adults classified by medical staff as "Level 1 trauma"; (6) adults deemed unable to provide informed consent (e.g. intoxication, mental incompetence, under guardianship); (7) patients treated in the ED for suicide attempts and sexual assault; (8) patients meeting past year drug abuse/dependence criteria; and (9) patients who have been in treatment for alcohol or other drug abuse/dependence in the previous year.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 686 (Actual)
Dates: Start 2005-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
receipt of assessment | 3 and 6 months post-baseline
treatment entry | 3 and 6 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frederic C Blow, PhD, Principal Investigator — University of Michigan
Locations (1):
- Hurley Medical Center, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No